CLINICAL TRIAL: NCT05663255
Title: Is Effectiveness of CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) Modulators Impacted by Co-therapy? A Population-based Comparative Effectiveness Study Using Data From French Cystic Fibrosis Registry Linked to French National Healthcare Insurance Database
Brief Title: Effectiveness of CFTR Modulators According to Co-therapy
Acronym: MODUCO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0066
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CFTR modulators; co-therapy; SNDS
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin; dornase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Patients treated with CFTR modulator with at least the discontinuation of one respiratory co-therapy (azithromycin, RhDNase, or inhaled antibiotics) during the year of initiation (A0) of CFTR modulator.
  Interventions: Drug: Discontinuation of respiratory co-therapy (azithromycin, RhDNase, or inhaled antibiotics)
- Control group: Patients treated with CFTR modulator without any discontinuation of respiratory co-therapy (azithromycin, RhDNase, inhaled antibiotics) during the year of initiation (A0) of CFTR modulator.

INTERVENTIONS:
Drug: Discontinuation of respiratory co-therapy (azithromycin, RhDNase, or inhaled antibiotics) — Discontinuation or reduction of at least one respiratory co-therapy (azithromycin, RhDNase, or inhaled antibiotics)
  Groups: Exposed group

SUMMARY:
Unless CFTR modulators are highly effective, the introduction of CFTR (Cystic fibrosis transmembrane conductance regulator) modulators could lead to concomitant reduction or discontinuation of respiratory co-therapies in real-life. Such reduction/discontinuation of respiratory co-therapies could lead to an overall decrease of the effectiveness of CF care.

MODUCO study aims: 1) to compare the clinical effectiveness on lung function and pulmonary exacerbation of CFTR modulator during the year of initiation, according to level of co-therapy among CF patients; 2) to describe the nature and level of respiratory co-therapies (azithromycin, RhDNase, inhaled antibiotics) in the year before the initiation of CFTR modulator; 3) to describe the changes in respiratory co-therapies during the first and the second year following the initiation of CFTR modulator and compare between the two CFTR modulators; 4) to describe adherence to CFTR modulator during the first and the second year following its initiation; 5) to study the association between the nature of respiratory co-therapies and adherence to CFTR modulator during the first and the second year following its initiation.

A national population-based comparative effectiveness study will be conducted, based on retrospective analysis of clinical and prescription data of the French CF registry linked with the French national health data system (SNDS).

ELIGIBILITY:
Inclusion Criteria:

* - CF patients aged 6 years and more,
* Treated at least 6 months by ivacaftor or lumacaftor/ivacaftor or elexacaftor/tezacaftor/ivacaftor,
* Included in the French CF registry,
* For whom probabilistic matching with the SNDS database has succeeded.

Exclusion Criteria:

* none

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Exhaustive on the recruitment of the all french CF patients meeting with eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1990 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung function | two years
  Change in the best forced expiratory volume in 1 second (FEV1) % predicted, measured during the year (A+1) compared to the year of initiation (A0) of CFTR modulator. The best FEV1 of the year is collected annually in the French CF Registry.